CLINICAL TRIAL: NCT03950154
Title: Phase III Clinical Study of PD-1 Monoclonal Antibody-activated Autologous Peripheral Blood T-lymphocyte (PD1-T) Combined With XELOX and Bevacizumab in the First-line Treatment of Recurrent and Metastatic Colorectal Cancer
Brief Title: Study of Chemotherapy Combination With Autologous Cell Immunotherapy in the Recurrent and Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2019-023-01
Record Dates: First submitted 2019-04-28; First posted 2019-05-15 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer
Keywords: effcet; safety
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Bevacizumab & Oxaliplatin & Capecitabine & PD1-T cells
  Bevacizumab, 7.5mg/kg, intravenous infusion, d1; Oxaliplatin, 130mg/m2, intravenous infusion, d1; Capecitabine, 1g/m2, oral administration, d1-14; PD1-T cells, 1x10^10 (10 billion), intravenous infusion, d17; Q3W, 6 cycles. After 6 cycles, Bevacizumab, 7.5mg/kg, intravenous infusion, d1; Capecitabine, 1g/m2, oral administration, d1-14; Q3W, maintenance treatment.
  Interventions: Drug: Bevacizumab Injection [Avastin]; Drug: Oxaliplatin; Drug: Capecitabine; Biological: PD1-T cells
- Arm 2: Control (Active Comparator): Bevacizumab & Oxaliplatin & Capecitabine
  Bevacizumab, 7.5mg/kg, intravenous infusion, d1; Oxaliplatin, 130mg/m2, intravenous infusion, d1; Capecitabine, 1g/m2, oral administration, d1-14; Q3W, 6 cycles. After 6 cycles, Bevacizumab, 7.5mg/kg, intravenous infusion, d1; Capecitabine, 1g/m2, oral administration, d1-14; Q3W, maintenance treatment.
  Interventions: Drug: Bevacizumab Injection [Avastin]; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Bevacizumab Injection [Avastin] — Bevacizumab injection
  Other Names: Avastin
Drug: Oxaliplatin — Oxaliplatin injection
Drug: Capecitabine — Capecitabine oral agent
Biological: PD1-T cells — PD1-T cells injection
  Other Names: PD-1 monoclonal antibody-activated peripheral blood T-lymphocyte
  Arms: Arm 1

SUMMARY:
This study evaluates the effect and safty of PD-1 monoclonal antibody-activated autologous peripheral blood lymphocyte (PD1-T) combined with XELOX and bevacizumab in the first-line treatment of recurrent and metastatic colorectal cancer. Half of participants receive PD1-T combined with XELOX and bevacizumab, while the other half will receive XELOX and bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

Subjects who must meet all the following criteria should be selected:

1. Agreeing to participate in this study and signing a written informed consent.
2. Male or female,from 18 to 75 years (including 18 and 75 years).
3. The life expectancy is longer than 3 months and can be followed up.
4. Patients with metastatic colorectal cancer whose condition has progressed after operation or could not receive radical surgery at initial treatment, will be confirmed by histological /cytological and imaging examinations. According to RECIST 1.1 standard, there will be at least one measurable lesion.
5. Bevacizumab, oxaliplatin and capecitabine were not used at least 6 months before the first administration of the drug in the patients with metastatic colorectal cancer whose condition has progressed after operation.
6. ECOG score will be 0 or 1 within 7 days before randomization.
7. Within 14 days before the start of treatment, the results of laboratory test of blood routine, liver, kidney function and hormone levels must be met the following criteria:

   White blood cells: more than 3.0 × 109/L; Platelets: more than 100 × 109/L; Neutrophils: more than 1.5 × 109/L; Hemoglobin: more than 80g/L; Serum glutamate pyruvate transaminase: less than 2.5 folds of the upper normal limit (ULN); Serum glutamic-oxal (o) acetic transaminase: less than 2.5 × ULN; Serum bilirubin: less than 1.25 × ULN; Serum creatinine: less than 1.25 × ULN. Cortisol and thyroid function will be in the normal range.
8. The toxicity and side effects of previous chemotherapy will must be alleviated to grade 1 or below (except hair loss).If the subjects received major surgical treatment or radiotherapy of > 30 Gy, they must recover from the toxicity or complications of these interventions, that is, they can be enrolled after 6 months.
9. Female subjects must take effective contraceptive measures throughout the study period; serum or urine pregnancy test results must be negative during screening and the whole study period.
10. Male subjects should take effective contraceptive measures from the beginning of treatment to within 6 months after the end of treatment.

Exclusion Criteria:

Subjects who meet any of the following criteria could not participate in this study:

1. Bevacizumab or oxaliplatin or capecitabine were used within 6 months before the first use of the study drug.
2. Patients received major surgery or local radiotherapy of more than 30 Gy within six months before the first use of the drug; received local radiofrequency, ablation, cryotherapy or radiotherapy of 30 Gy or less within one month before the first use of the drug; or received anti-tumor monoclonal antibody (mAb), chemotherapy and targeted small molecule therapy within one month before the first use of the drug. Patients with metastases who can undergo radical surgery.
3. Other malignant tumors needed treatment within five years.
4. Allogeneic tissue/organ transplantation.
5. Participating in research drug therapy within 4 weeks before the first administration of the trial.
6. Systemic glucocorticoid therapy or any other form of immunosuppressive therapy (except glucocorticoid preconditioned with docetaxel) is being administered within 3 days before the first administration of the experimental therapy.
7. Previous treatment with PD-1/PD-L1 antibodies.
8. Over the past two years, patients with active autoimmune diseases requiring systemic treatment, such as the use of corticosteroids, or immunosuppressants. Substitution therapy (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary dysfunction) is not a systemic treatment.
9. Having bleeding tendency, high risk of bleeding or coagulation dysfunction, having a history of thrombosis within 6 months and/or hemoptysis within 3 months; being treated with full oral and/or parenteral anticoagulants and thrombolysis agents (preventive use of anticoagulants is permitted); having used aspirin or other non-steroidal anti-inflammatory drugs that inhibit platelet function within 10 days; / MR imaging showed that the tumors surrounded or invaded the large vessel lumen.
10. Patients with congenital or acquired immunodeficiency (e.g. HIV-infected persons), active hepatitis B (HBV-DNA > 10^3 copies/ml) or hepatitis C (hepatitis C antibody positive), and HCV-RNA higher than the detection limit of the analytical method.
11. Poorly controlled hypertension (systolic pressure 150 mmHg and/or diastolic pressure 100 mmHg), previous hypertension crisis and hypertensive encephalopathy, and severe cerebrovascular diseases.
12. Non-healing wounds, active peptic ulcer, tracheoesophageal fistula, gastrointestinal perforation and abdominal abscess within 6 months.
13. Subjects with active central nervous system (CNS) metastases and/or cancerous meningitis.
14. Patients with active infections requiring systemic intravenous therapy.
15. Mental illness or other illnesses, such as uncontrollable heart disease or pulmonary disease, diabetes, etc.
16. Subjects who are known to be allergic to any of the constituents of the drug being studied.
17. Subjects with a recent history of drug abuse (including alcohol) within one year.
18. Compliance is poor and can not cooperate with clinical research.
19. Female subjects who are pregnant or breastfeeding, or who are expected to be pregnant during the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  PFS will be calculated from initiation of treat- ment until first progression, and patients alive in stable state will be censored at the time of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Xiubao Ren, MD. PhD., Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Pan QZ, Zhao JJ, Liu L, Zhang DS, Wang LP, Hu WW, Weng DS, Xu X, Li YZ, Tang Y, Zhang WH, Li JY, Zheng X, Wang QJ, Li YQ, Xiang T, Zhou L, Yang SN, Wu C, Huang RX, He J, Du WJ, Chen LJ, Wu YN, Xu B, Shen Q, Zhang Y, Jiang JT, Ren XB, Xia JC. XELOX (capecitabine plus oxaliplatin) plus bevacizumab (anti-VEGF-A antibody) with or without adoptive cell immunotherapy in the treatment of patients with previously untreated metastatic colorectal cancer: a multicenter, open-label, randomized, controlled, phase 3 trial. Signal Transduct Target Ther. 2024 Apr 3;9(1):79. doi: 10.1038/s41392-024-01788-2. PMID 38565886